CLINICAL TRIAL: NCT06633380
Title: Alternative Physical Activity Strategies for Breast and Prostate Cancer Survivors
Brief Title: Alternative Physical Activity Strategies for Breast Cancer Survivors
Acronym: PACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Amy Kirkham, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB #44269
Record Dates: First submitted 2024-09-13; First posted 2024-10-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Insulin Resistance; Cardiometabolic Risk Factors
Keywords: Physical Activity; Hormone Therapy; Glycemic Control
MeSH Terms: conditions — Breast Neoplasms; Insulin Resistance; Motor Activity

STUDY DESIGN:
Intervention Model Description: 5-arm randomized crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard Physical Activity - Fasted (Experimental): Participants will perform 30 minutes of walking at a self-selected pace 15 minutes prior to consumption of first meal in the morning (including cream/sugar/milk in coffee or tea).
  Interventions: Behavioral: Standard Physical Activity - Fasted
- Standard Physical Activity - Post-Meal (Experimental): Participants will perform 30 minutes of walking at a self-selected pace 30 minutes after the start of the first meal in the morning.
  Interventions: Behavioral: Standard Physical Activity - Post-Meal
- Dispersed Physical Activity (Experimental): Participants will perform 10 minutes of walking at a self-selected pace 30 minutes after the start of each main meal throughout the day (i.e., three bouts total).
  Interventions: Behavioral: Dispersed Physical Activity
- Physical Activity Snacks (Experimental): Participants will perform 2 minutes of walking or marching on the spot at a self-selected pace every 30 minutes throughout the day for 7.5 waking hours.
  Interventions: Behavioral: Physical Activity Snacks
- Muscle Strengthening (Experimental): Participants will perform 30 minutes of muscle strengthening exercises targeting the major muscle groups of the whole body performed by following along with a video, to start 30 minutes after the start of the first meal in the morning.
  Interventions: Behavioral: Muscle Strengthening

INTERVENTIONS:
Behavioral: Standard Physical Activity - Fasted — 30 minutes of walking at a self-selected pace that they must have completed 15 minutes prior to consumption of first meal in the morning.
  Arms: Standard Physical Activity - Fasted
Behavioral: Standard Physical Activity - Post-Meal — 30 minutes of walking at a self-selected pace to start 30 minutes after the start of the first meal in the morning.
  Arms: Standard Physical Activity - Post-Meal
Behavioral: Dispersed Physical Activity — 10 minutes of walking at a self-selected pace to start 30 minutes after the start of each main meal throughout the day (i.e., three bouts total).
  Arms: Dispersed Physical Activity
Behavioral: Physical Activity Snacks — 2 minutes of walking or marching on the spot at a self-selected pace every 30 minutes throughout the day for 7.5 waking hours.
  Arms: Physical Activity Snacks
Behavioral: Muscle Strengthening — 30 minutes of muscle strengthening exercises targeting the major muscle groups of the whole body, to start 30 minutes after the start of the first meal in the morning.
  Arms: Muscle Strengthening

SUMMARY:
The primary aim of this study is to compare the acute glycemic effects of two novel, alternative physical activity (PA) strategies (dispersed post-meal PA, PA snacks) to a no PA condition and to exercise sessions representing the PA guidelines (standard 30-minute walking bout performed under fasting and under postprandial conditions and a standard 30-minute resistance training session) among sedentary breast cancer survivors who are currently receiving hormone therapies and age- and BMI-matched postmenopausal women without a history of cancer. The secondary aim is to determine whether the alternative PA strategies are acceptable and feasible in the free-living setting. An exploratory aim is to determine whether the outcomes differ between women with and without a history of breast cancer and use of aromatase inhibitors.

The investigators hypothesize that:

1. Dispersed PA and PA snacks will result in greater reductions in 24-hour glucose and postprandial glucose compared to the no-PA baseline and similar reductions to a standard 30-minute bouts of walking;
2. The alternative PA strategies will be more feasible and have greater acceptability by cancer survivors compared to the standard 30-minute bout of walking or resistance training; and
3. The different PA strategies will have similar effects on glycemic outcomes for both breast cancer survivors and cancer-free controls. The resistance exercise session is an exploratory trial as the effects of it on acute glycemic control are understudied.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal biological females diagnosed with stage I, II, or III breast cancer and currently using aromatase inhibitors (AI) for at least 3 months prior to start of study participation
* All participants must meet the following criteria:

  * Body mass index equal to or greater than 25 kg/m^2.
  * Self-report consuming three main meals daily.
  * Self-report as being sedentary (i.e., less than 30 minutes/week of moderate-to-vigorous aerobic physical activity and less than twice/week muscle strengthening of major muscle groups in the last three months.

Exclusion Criteria:

* If unable or unwilling to receive medical clearance by a physician after being screened for major signs or symptoms of cardiovascular diseases, diabetes, or renal disease and safety to initiate exercise.

  * Major signs or symptoms of cardiovascular diseases, diabetes, or renal disease are taken from the American College of Sports Medicine's Guidelines for Exercise Testing and Prescription 11th edition Table 2.1. They include pain or discomfort in the chest, neck, jaw, arms with rest or exercise, shortness of breath at rest or with mild exertion, dizziness or syncope, ankle edema, palpitations or tachycardia, intermittent claudication, known heart murmur, and unusual fatigue with usual activities.
  * Safety to initiate exercise will be screened using the Get Active Questionnaire, which is the Canadian Society of Exercise Physiology's endorsed evidence-based pre-screening tool.
* Using drugs for diabetes management (e.g., exogenous insulin, Ozempic, metformin, etc.) or actively losing weight (i.e., >5 kg weight loss in past 3 months) from drugs or other reasons
* Report any injury or other reason for not feeling capable of completing a 30 minute continuous walk or muscle strengthening exercise
* Unable to access an Ontario Lifelabs location for an overnight fasted blood draw
* Do not have a smartphone compatible with the applications required to collect data.
* Cannot read and understand the consent form or communicate in English.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
24-hour glucose incremental area under the curve (iAUC) | Baseline, 24 hours of each intervention day
  Assessed for each single-day intervention using a continuous glucose monitor from 8:00 am to the intervention day to 8:00 am the following morning.

SECONDARY OUTCOMES:
24-hour mean glucose | Baseline, 24 hours of each intervention day
  Assessed for each single-day intervention using a continuous glucose monitor from 8:00 am to the intervention day to 8:00 am the following morning.
Postprandial iAUC | Baseline, 24 hours of each intervention day
  Assessed for each single-day intervention using a continuous glucose monitor for two hours following each meal.
Peak postprandial glucose | Baseline, 24 hours of each intervention day
  Assessed as the highest glucose concentration during the 2 hours following each meal using a continuous glucose monitor.
Daytime glucose concentration | Baseline, 24 hours of each intervention day
  Assessed for each single-day intervention using a continuous glucose monitor from 6:00 am to 12:00 am on the intervention day.
Nocturnal glucose concentration | Baseline, 24 hours of each intervention day
  Assessed for each single-day intervention using a continuous glucose monitor from 12:00 am to 6:00 am on the intervention day.
Time in hypoglycemia | Baseline, 24 hours of each intervention day
  Assessed as the number of hours with glucose less than 3.9 mmol/L using a continuous glucose monitor.
Time in hyperglycemia | Baseline, 24 hours of each intervention day
  Assessed as the number of hours with glucose greater than 10 mmol/L using a continuous glucose monitor.
Indices of glycemic variability | Baseline, 24 hours of each intervention day
  Indices include standard deviation, coefficient of variation, mean amplitude of glycemic excursion, and continuous overall net glycemic action
Participant acceptability | 24 hours of each intervention day
  Acceptability related to participants' experience with each single-day intervention will be assessed using a researcher-developed questionnaire at the end of each intervention day. Seven items use a 5-point Likert scale with responses ranging from "Strongly Disagree" to "Strongly Agree", while four items ask about participant confidence with responses ranging from 0 ("Not Confident") to 10 ("Very Confident). A higher total score indicates the intervention is more acceptable to the participant.
Participant enjoyment | 24 hours of each intervention day
  Enjoyment related to participants' experience with each single-day intervention will be assessed using the short form of the Physical Activity Enjoyment Scale at the end of each intervention day, consisting of 8 items each scored on a 7-point Likert scale, with the total score ranging from 8 to 56, and a higher total score indicating greater enjoyment.

OTHER OUTCOMES:
Physical activity | 24 hours of each intervention day
  Participants will be asked to wear a Garmin smartwatch for the duration of the study to track completion of physical activity bouts and heart rate during each bout for each single-day intervention
Systolic and Diastolic Blood Pressure | Baseline
  Measured as the average of the last 5 of 6 systolic and diastolic blood pressure measurements using an automatic blood pressure device.
Waist circumference | Baseline
  Circumference of the waist measured using an inelastic tape
Body mass index (BMI) | Baseline
  Calculated using self-reported body weight and height.
Fasting glucose | Baseline
  Analyzed from fasted (overnight, 12 hours) venipuncture performed and processed at any Lifelabs location of participant's choice.
Fasting insulin | Baseline
  Analyzed from fasted (overnight, 12 hours) venipuncture performed and processed at any Lifelabs location of participant's choice.
Lipid profile: HDL, LDL, total cholesterol, triglycerides | Baseline
  Analyzed from fasted (overnight, 12 hours) venipuncture performed and processed at any Lifelabs location of participant's choice.
Hemoglobin A1c | Baseline
  Analyzed from fasted (overnight, 12 hours) venipuncture performed and processed at any Lifelabs location of participant's choice.
Metabolic syndrome | Baseline
  Determined based on standardized criteria using previously specified outcomes.
Framingham 10-year cardiovascular disease risk score | Baseline
  Calculated via a standardized scoring algorithm using previously specified outcomes, with total scores ranging from less than -3 (indicating <1% 10-year risk of cardiovascular disease) to more than 21 (indicating >30% 10-year risk of cardiovascular disease).
Dietary intake | Baseline
  Various components of dietary intake including macronutrients and micronutrients will be assessed through 1-day food record on a weekday collected using ASA-24 online system.
Perceived stress | Prior to start of each intervention
  Assessed using a researcher-developed visual analog scale (0-100, with a higher value indicating greater perceived stress) at the start of each intervention day.
Muscle soreness | Prior to start of each intervention
  Assessed using a researcher-developed visual analog scale (0-100, with a higher value indicating greater muscle soreness) at the start of each intervention day.
Sleep quantity and quality | Baseline, 24 hours of each intervention day
  Measured via Garmin smartwatch for the total sleep duration and efficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- Remote Ontario-wide, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No